CLINICAL TRIAL: NCT03555500
Title: Fasting Versus Non-fasting Prior To Elective Cardiac Catheterization
Brief Title: Fasting or Non Fasting for Cardiac Catheterization
Acronym: FANPRECC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blackpool Victoria Hospital (Other)
Responsible Party: Principal Investigator, Hesham Abdelaziz, Interventional Cardiologist, Blackpool Victoria Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 215149
Record Dates: First submitted 2018-05-10; First posted 2018-06-13 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Fasting; Cardiac Catheterization
Keywords: Fasting; Non fasting; Cardiac catheterization
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting Group (No Intervention): Clear fluids up to the time of the procedure and no food for at least 2 hours before the procedure.
- Non fasting group (Experimental): Clear fluids and food up to the time of the procedure.
  Interventions: Other: Non fasting

INTERVENTIONS:
Other: Non fasting — Non fasting group is allowed for clear fluids and food up to the time of the procedure.
  Arms: Non fasting group

SUMMARY:
The current practice of fasting before cardiac catheterization is not based on any studies. If the procedure is to be delayed ( which is common due to busy catheterization lab), this could result in patient's dis-satisfaction and hypoglycemia. Occasionally, cancellation occur because patients are found to be non fasting ( not following the current protocol). The old data of fasting was extrapolated from procedure done under general anesthesia. Now days, cardiac catheterization is always done under local anesthesia and mild sedation. As a matter of fact, emergency cardiac catheterization done for heart attack patients carries more risk than elective one , and are still done without fasting with no reported complication rate like lung aspiration . The highest level of evidence to change the current practice comes from randomized control study. This study has been designed to challenge the current practice. The patients will be divided into 2 groups:

* Fasting group (current practice): Clear fluids up to the time of the procedure and no food for at least 2 hours before the procedure.
* Non Fasting Group: clear fluids and food and up to the time of the procedure

The investigators' aim is to show that there is no difference with regards to potential complications between fasting (current practice) and non fasting (new practice) groups of patients with less incidence of hypoglycemia and hypotension in non fasting group. In addition, The investigators believe that patient satisfaction will be improved if patients are allowed to eat freely before the procedure and the catheter lab working ability will be maximized as the list can be filled promptly with patient on the waiting list (as fasting is no longer required) if a previously booked patient has to be cancelled in the last minute improving patient experience along with the associated financial benefits.

DETAILED DESCRIPTION:
All patients to be admitted electively for coronary angiography or angioplasty will be given the opportunity to participate. An invitation letter together with patient information leaflet outlining the study will be sent along with the pre-procedure appointment letter to give the patient time to read and think about the study. Once at pre-procedure assessment clinic, the study will be explained further including potential risks and intended outcome and patients concerns will be addressed. Patient will be given the opportunity either to take part in the study or abstain and follow the standard procedure. If the patient agrees then they will sign the consent form and then be randomised in a 1:1 ratio to either the fasting or non-fasting group and be allocated a patient identification number. This will be done at the pre-procedure assessment clinic.

1. Fasting group (current practice): Clear fluids up to the time of the procedure and no food for at least 2 hours before the procedure.
2. Non Fasting Group: Clear fluids and food up to the time of the procedure. The pre procedure preparation will then be documented in the notes. Intention to treat analysis will be used to avoid the effects of crossover and dropout providing unbiased comparisons among the treatment groups.

Finally once the patient is ready for discharge they will be asked to complete an anonymous questionnaire relating to their experience and satisfaction.All patients will be contacted by phone on day 30 or the nearest working day thereafter to ensure no chest infections

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years undergoing elective coronary angiography or angioplasty procedures

Exclusion Criteria:

* Patient choice
* Other cardiac procedures such as EP studies, pacing, structural heart disease intervention
* Emergency PPCI
* Patients already admitted in the hospital with UA / NSTEMI
* Patients unable to give informed consent (vulnerable group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-03-10 (Estimated)

PRIMARY OUTCOMES:
Composite incidence of nausea, vomiting, abdominal pain, emergency intubation and aspiration | 8 hours
  The incidence of any of nausea, vomiting, abdominal pain aspiration or emergency intubation during the procedure and up to 8 hours will be recorded.

SECONDARY OUTCOMES:
Incidence of hypoglycaemia | 1 hour
  Drop of Blood sugar < 3.6 mmol/l as assessed by finger prick test before the procedure.
Incidence of hypotension | 1 hour
  Drop of SBP<90 mmHg and /or DBP<60 mmHg as measured by manual sphygmomanometer before the procedure.
Patient satisfaction | 1 hour
  A questionnaire given to the patient after the procedure to assess their experience , symptoms and overall satisfaction with regard to the procedure. The questionnaire include a preset of yes/no question including feeling hungry, thirsty or lethargic before the procedure, feeling headache, nausea or vomited during or up to 1 hour after the procedure. then a final overall satisfaction score about the procedure today from 1- 5, with 1 being not satisfied and 5 being extremely satisfied.
chest infection | At 30 days
  All patients will be contacted or reviewed in clinic to assess for chest infection

CONTACTS AND LOCATIONS:
Overall Officials: Hesham abdelaziz, Ph.D, Principal Investigator — Blackpool Victoria Hospital -UK
Locations (1):
- Blackpool Victoria Hospital, Blackpool, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godwin SA, Burton JH, Gerardo CJ, Hatten BW, Mace SE, Silvers SM, Fesmire FM; American College of Emergency Physicians. Clinical policy: procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2014 Feb;63(2):247-58.e18. doi: 10.1016/j.annemergmed.2013.10.015. PMID 24438649
- [Background] Association of Anaesthetists of Great Britain and Ireland; Farling PA, Flynn PA, Darwent G, De Wilde J, Grainger D, King S, McBrien ME, Menon DK, Ridgway JP, Sury M, Thornton J, Wilson SR. Safety in magnetic resonance units: an update. Anaesthesia. 2010 Jul;65(7):766-70. doi: 10.1111/j.1365-2044.2010.06377.x. PMID 20642539
- [Background] Rosengarten J, Ozkor M, Knight C. Fasting and cardiac catheterization should we be following the evidence. Controversies and Consensus in Imaging and Intervention (C2I2) 2007;V5:22-3
- [Background] Brady M, Kinn S, Stuart P. Preoperative fasting for adults to prevent perioperative complications. Cochrane Database Syst Rev. 2003;(4):CD004423. doi: 10.1002/14651858.CD004423. PMID 14584013
- [Result] Kwon OK, Oh CW, Park H, Bang JS, Bae HJ, Han MK, Park SH, Han MH, Kang HS, Park SK, Whang G, Kim BC, Jin SC. Is fasting necessary for elective cerebral angiography? AJNR Am J Neuroradiol. 2011 May;32(5):908-10. doi: 10.3174/ajnr.A2408. Epub 2011 Mar 17. PMID 21415144
- [Result] Hamid T, Aleem Q, Lau Y, Singh R, McDonald J, Macdonald JE, Sastry S, Arya S, Bainbridge A, Mudawi T, Balachandran K. Pre-procedural fasting for coronary interventions: is it time to change practice? Heart. 2014 Apr;100(8):658-61. doi: 10.1136/heartjnl-2013-305289. Epub 2014 Feb 12. PMID 24522621

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT03555500/Prot_SAP_000.pdf